CLINICAL TRIAL: NCT00959023
Title: UK Genetic Prostate Cancer Study
Brief Title: Study of Blood and Tumor Samples From Men With an Inherited Risk of Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000636371; ICR-UKGPCS; EU-20909
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: medical chart review
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify genes related to cancer.

PURPOSE: This clinical trial is studying blood and tumor samples from men with an inherited risk of prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To find genes that predispose to prostate cancer (using genetic linkage and other molecular biology techniques).
* To determine if genes that predispose to prostate cancer are associated with disease and treatment parameters.
* To determine if genes that predispose to prostate cancer are associated with environmental factors.
* To estimate the percentage of prostate cancer patients who have a positive family history of the disease.
* To estimate the relative risk of developing prostate cancer in a currently unaffected member of a prostate cancer family.
* To ascertain whether relatives of prostate cancer patients are at increased risk of developing cancers other than prostate cancer.
* To build up a large blood and tumor (both fresh and preserved) bank from patients with prostate cancer to identify prostate cancer predisposition gene(s), determine the prevalence and penetrance of prostate cancer predisposition genes in prostate cancer patients, correlate changes in prostate cancer predisposition gene(s) with disease and treatment parameters by matching with clinical data from clinical databases already held as part of the medical record on these patients, and correlate changes in prostate cancer predisposition gene(s) with environmental factors collected by questionnaire from these patients.
* To use the blood and tumor bank for marker studies (DNA, RNA, serum, plasma, protein, and other molecules) to define the role of these markers in disease prediction and progression.
* To develop microarrays from prostate cancers to determine their genetic profile and correlate this with prostate cancer genetic predisposition genes.
* To collect tissue from other unaffected and affected members of the family in cases where a genetic alteration is found, in order to ascertain whether this alteration is associated with disease risk.
* To collect tissue samples from unaffected family members who show an interest in taking part in the study.

OUTLINE: Patients are assessed by a family history and epidemiology questionnaire and undergo a medical record review.

Patients and relatives with prostate cancer may undergo blood sample collection for genetic analysis of prostate cancer predisposition genes and measurement of markers of associations with genetic changes associated with prostate cancer. Blood and tumor samples are stored for future studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of prostate cancer meeting any of the following criteria:

    * Attending prostate clinics at The Royal Marsden NHS Foundation Trust

      * Any age at diagnosis
    * Not attending prostate clinics at The Royal Marsden NHS Foundation Trust, meeting 1 of the following criteria:

      * No older than 60 years at diagnosis
      * Diagnosis in two relatives where one is ≤ 65 years at diagnosis
      * At any age in a cluster with 3 or more cases
  * Any unaffected male relatives of men who are already taking part in the study

PATIENT CHARACTERISTICS:

* Able to understand the information sheet and give informed consent
* No man who is too ill to take part

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21000 (Estimated)
Dates: Start 1993-06

PRIMARY OUTCOMES:
Prostate cancer (PC) predisposition (PCP) genes

SECONDARY OUTCOMES:
Association of PCP genes with disease and treatment parameters
Association of PCP with environmental factors
Family history of PC
Relative risk of developing PC
Increased risk relatives of PC patients are to develop cancers other than PC
Markers of PC that are associated with PCP genes
Specific tumor genetic profile correlated with PCP genes

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Eeles, PhD, FRCR, FRCP, FMed Sci, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (135):
- United Kingdom (135):
  - William Harvey Hospital, Ashford-Kent, England
  - Tameside General Hospital, Ashton-under-Lyne, England
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - North Devon District Hospital, Barnstaple, England
  - Furness General Hospital, Barrow in Furness, England
  - Basildon University Hospital, Basildon, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Royal United Hospital, Bath, England
  - Primrose Centre at Bedford Hospitals NHS Trust, Bedford, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - City Hospital - Birmingham, Birmingham, England
  - Good Hope Hospital, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Royal Blackburn Hospital, Blackburn, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Pilgrim Hospital, Boston, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Southmead Hospital, Bristol, England
  - Frenchay Hospital, Bristol, England
  - Bristol Royal Infirmary, Bristol, England
  - Broomfield Hospital, Broomfield, England
  - Burnley General Hospital, Burnley, England
  - Queen's Hospital, Burton-on-Trent, England
  - Addenbrooke's Hospital, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - St. Helier Hospital, Carshalton, England
  - Countess of Chester Hospital, Chester, England
  - Colchester General Hospital, Colchester, England
  - Castle Hill Hospital, Cottingham, England
  - Walsgrave Hospital, Coventry, England
  - Mid Cheshire Hospitals Trust- Leighton Hopsital, Crewe, England
  - Mayday University Hospital, Croydon, England
  - Darent Valley Hospital, Dartford Kent, England
  - Derbyshire Royal Infirmary, Derby, England
  - Royal Derby Hospital, Derby, England
  - Dorset County Hospital, Dorchester, England
  - Russells Hall Hospital, Dudley, England
  - Eastbourne District General Hospital, Eastbourne, England
  - Birmingham Women's Hospital, Edgbaston, England
  - Epsom General Hospital, Epsom, Surrey, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Royal Bolton Hospital, Farnworth, England
  - Frimley Park Hospital, Frimley, England
  - Grantham and District Hospital, Grantham, Lincolnshire, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - Harrogate District Hospital, Harrogate, England
  - Wycombe General Hospital, High Wycombe, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Kidderminster Hospital, Kidderminster Worcestershire, England
  - Royal Albert Edward Infirmary, Lancanshire, England
  - Royal Lancaster Infirmary, Lancaster, England
  - Leeds General Infirmary, Leeds, England
  - Cookridge Hospital, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Leicester General Hospital, Leicester, England
  - Lincoln County Hospital, Lincoln, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Royal London Hospital, London, England
  - Whipps Cross Hospital, London, England
  - Saint Bartholomew's Hospital, London, England
  - Guy's Hospital, London, England
  - Hammersmith Hospital, London, England
  - Middlesex Hospital, London, England
  - St. Mary's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Macclesfield District General Hospital, Macclesfield, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Milton Keynes General Hospital, Milton Keynes, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham City Hospital, Nottingham, England
  - Kings Mill Hospital, Nottinghamshire, England
  - George Eliot Hospital, Nuneaton, England
  - Churchill Hospital, Oxford, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - Queens Hospital, Romford, England
  - Conquest Hospital, Saint Leonards-on-Sea, England
  - Hope Hospital, Salford, England
  - Salisbury District Hospital, Salisbury, England
  - Scarborough General Hospital, Scarborough, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Solihull Hospital, Solihull, England
  - Southampton General Hospital, Southampton, England
  - Southport and Formby District General Hospital, Southport, England
  - Staffordshire General Hospital, Stafford, England
  - Lister Hospital, Stevenage, England
  - Stirling Royal Infirmary, Stirling, England
  - Stepping Hill Hospital, Stockport, England
  - Kingston Hospital, Surrey, England
  - East Surrey Hospital, Surrey, England
  - Royal Marsden - Surrey, Sutton, England
  - Great Western Hospital, Swindon, England
  - Taunton and Somerset Hospital, Taunton, England
  - Torbay Hospital, Torquay, England
  - Hillingdon Hospital, Uxbridge, England
  - Warwick Hospital, Warwick, England
  - Sandwell General Hospital, West Bromwich, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - New Cross Hospital, Wolverhampton, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil, England
  - Cancer Care Centre at York Hospital, York, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Downe Hospital, Downpatrick, Northern Ireland
  - Altnagelvin Area Hospital, Londonderry, Northern Ireland
  - Craigavon Area Hospital, Portadown, Craigavon, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ayr Hospital, Ayr, Scotland
  - Falkirk and District Royal Infirmary, Falkirk, Scotland
  - Western Infirmary, Glasgow, Scotland
  - Pinderfields General Hospital, Wakefield, Scotland
  - Princess of Wales Hospital, Bridgend, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - University Hospital of Wales, Cardiff, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Singleton Hospital, Swansea, Wales
  - Queen Victoria Hospital, Morecambe
  - Edith Cavell Hospital, Peterborough
  - Southlands Hospital, Shoreham-by-Sea
  - Princess Anne Hospital, Southampton